CLINICAL TRIAL: NCT01210729
Title: Mechanical Recanalization With Flow Restoration in Acute Ischemic Stroke (ReFlow Study)
Brief Title: Mechanical Recanalization With Flow Restoration in Acute Ischemic Stroke
Acronym: ReFlow
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universität des Saarlandes (Other)
Responsible Party: Prof. Wolfgang Reith, Department of diagnostic and interventional Neuroradiology, Saarland University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ReFlow01
Record Dates: First submitted 2010-09-27; First posted 2010-09-28 (Estimated); Last update posted 2011-12-02 (Estimated); Status verified 2010-09

CONDITIONS: Acute Stroke
Keywords: stroke; mechanical recanalization; self-expanding stent; Solitaire
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Solitaire FR, ev3 — Placement of the stent in the occluded vessel segment, withdrawal in its unfolded state.
  Other Names: device used: Solitaire FR, ev3, USA

SUMMARY:
The objective of this study is to collect data on the use of the SOLITAIR FR device for treatment of acute ischemic stroke with large artery occlusion i.e. to investigate, whether the application of SOLITAIR is a safe and feasible method for interventional recanalization of large vessels with favorable patient outcome in acute stroke therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-85 years
* Acute ischemic stroke with occlusion if ICA, MCA, VA or BA (TICI 0 or 1 flow) within the first 6 hours

Exclusion Criteria:

* Rapidly improving neurological signs
* NHISS>30 or coma
* Female patients, who are pregnant or lactating
* Use of warfarin anticoagulation with INR > 1.5
* Platelet count < 30,000
* Glucose < 50 mg/dL
* Life expectancy of less than 90 days
* Computed tomography (CT) or Magnetic Resonance Imaging (MRI) evidence of hemorrhage on presentation
* CT showing hypodensity on presentation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2010-09; Primary Completion 2011-11 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Overall frequency of favourable clinical outcome (modified Rankin Scale 0 to 2), and unfavourable clinical outcome or death (modified Rankin Scale 3 to 6) | Day 90

SECONDARY OUTCOMES:
Arterial recanalization of occluded target vessel measured by Thrombolysis in Cerebral Infarction (TICI)score of 2b or 3 following the use of the SOLITAIRE FR Device | Day 0
Excellent functional clinical outcome (modified Rankin Scale 0 or 1) | Day 90
All causes of mortality | Day 90
Proportion of patients with rapid neurological improvement (more than 4 points on the NIHSS) during the first 24 hours after treatment. | Day 1
Symptomatic intracranial haemorrhages up to 24 hours after treatment defined as homogeneous areas of haemorrhage, with or without mass effect or intraventricular extension with neurological deterioration | Day 1
Time between arterial puncture and Flow Restoration | Day 0
Time between arterial puncture and TICI 2b or 3 recanalization | Day 0
Number of SOLITAIRE device runs until recanalization | Day 0
Number of patients with and degree of stenosis in the treated artery 90 days after recanalization with SOLITAIRE | Day 90
Number of patients in which thrombus material was preserved | Day 0
Histological examination of the thrombus material in correlation with TICI 2b or 3 recanalization and favorable clinical outcome | Day 1
Overall frequency of modified Rankin Scale 0 to 2 at 30 days | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Reith, MD, Principal Investigator — Saarland University Hospital
Locations (1):
- Department of diagnostic and interventional Neuroradiology, Homburg, Saarland, Germany

REFERENCES:
- [Background] Papanagiotou P, Roth C, Walter S, Behnke S, Politi M, Fassbender K, Haass A, Reith W. Treatment of acute cerebral artery occlusion with a fully recoverable intracranial stent: a new technique. Circulation. 2010 Jun 15;121(23):2605-6. doi: 10.1161/CIRCULATIONAHA.110.948166. No abstract available. PMID 20547941
- [Background] Roth C, Papanagiotou P, Behnke S, Walter S, Haass A, Becker C, Fassbender K, Politi M, Korner H, Romann MS, Reith W. Stent-assisted mechanical recanalization for treatment of acute intracerebral artery occlusions. Stroke. 2010 Nov;41(11):2559-67. doi: 10.1161/STROKEAHA.110.592071. Epub 2010 Oct 14. PMID 20947848
- [Background] Papanagiotou P, Roth C, Walter S, Behnke S, Grunwald IQ, Viera J, Politi M, Korner H, Kostopoulos P, Haass A, Fassbender K, Reith W. Carotid artery stenting in acute stroke. J Am Coll Cardiol. 2011 Nov 29;58(23):2363-9. doi: 10.1016/j.jacc.2011.08.044. PMID 22115640
- [Background] Papanagiotou P, Roth C, Reith W. Letter by Papanagiotou et Al regarding article, "percutaneous vascular interventions for acute ischemic stroke". Stroke. 2011 Sep;42(9):e545; author reply e546. doi: 10.1161/STROKEAHA.111.620989. Epub 2011 Jul 14. No abstract available. PMID 21757666
- [Derived] Roth C, Reith W, Walter S, Behnke S, Kettner M, Viera J, Yilmaz U, Alexandrou M, Politi M, Kostopoulos P, Korner H, Krick C, Haass A, Fassbender K, Papanagiotou P. Mechanical recanalization with flow restoration in acute ischemic stroke: the ReFlow (mechanical recanalization with flow restoration in acute ischemic stroke) study. JACC Cardiovasc Interv. 2013 Apr;6(4):386-91. doi: 10.1016/j.jcin.2012.11.013. Epub 2013 Mar 20. PMID 23523460